CLINICAL TRIAL: NCT00481754
Title: Benign Reproductive Tissue Evaluation (BRTE) Study
Brief Title: Benign Reproductive Tissue Analysis for Endometrial Cancer Markers
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999906109; 06-C-N109; NCT00342680 (obsolete NCT alias)
Record Dates: First submitted 2007-06-01; First posted 2007-06-04 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Oophorectomy for Benign Reasons; Hysterectomy
Keywords: Endometrium; PTEN; Hormones; Carcinogenesis; Etiology; Tissue Evaluation; Questionnaire
MeSH Terms: conditions — Carcinogenesis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Females with ovarian cancer: Recruited from Magee Women's Hospital

SUMMARY:
Background:

* Endometrial cancer (cancer of the lining of the uterus) is the most common gynecologic cancer in the United States.
* Currently, there are no markers (components of blood and tissue that determine who might be at risk for developing cancer) for endometrial cancer.

Objectives:

-To see if women who are undergoing hysterectomy are willing to provide blood and tissue samples to help doctors identify markers that would indicate increased risk for developing endometrial cancer.

Eligibility:

-Women between 35 and 54 years of age who will undergo hysterectomy for a non-cancerous condition, such as uterine fibroids, uterine prolapse, abnormal uterine bleeding, and others at Magee-Women's Hospital in Pittsburgh, Penn.

Design:

* Patients' medical records are reviewed and patients complete a questionnaire including information on race and ethnic background, education, marital status, family history, height, weight, pregnancy history, smoking history, medication history, history about menstrual periods and menopausal symptoms.
* Patients provide blood and urine samples before surgery.
* A sample of fat tissue is removed during surgery in patients undergoing abdominal surgery.
* Tissue samples from the removed uterus (and ovaries if the ovaries are also removed) are collected and analyzed for markers for endometrial cancer.

DETAILED DESCRIPTION:
Our hypothesis is that silent molecular lesions, defined as molecular alterations

detectable in histologically normal endometrial, ovarian, and tubal tissues, represent markers of cancer risk. Incessant ovulation represents one of the most widely-recognized models to explain the pathogenesis of ovarian cancer, with women who have had a high number of lifetime ovulatory menstrual cycles being at increased cancer risk because of repeated ovulation-related injury to, and repair of, ovarian surface epithelium (OSE). This extremely delicate single layer of cells exfoliates easily on handling, with the majority of cells typically being lost in routine handling, when collected post-operatively. Furthermore, the identification of early stage ovarian cancer is uncommon, and the vast majority of ovarian cancers are not associated with recognizable precursors. The lack of effective techniques for collecting and studying OSE in the laboratory represents a major barrier to molecular studies designed to uncover the etiology and early pathogenesis of ovarian cancer. This proposal will develop a collection method for OSE, and demonstrate its utility for various molecular analyses. Recent evidence suggests that a subset of ovarian cancers may originate in the fallopian tubes. Therefore, we will pilot the collection of cells from the fallopian tubes. If successful, the collection of OSE and fallopian tube cells will provide the basis for larger studies aimed at identifying early molecular events in ovarian carcinogenesis.

In this pilot, we will collect endometrial and ovarian tissues (that would otherwise have been discarded without histopathologic examination) from 125 hysterectomy and/or unilateral or bilateral oophorectomy specimens obtained from women ages 18 and older who were operated on for benign indications. As an amendment to this active protocol, we propose demonstrating the feasibility of obtaining intra-operative cytobrushings of ovarian surface epithelial cells on 50 women to be accrued onto the study, which will include women having hysterectomy (or unilateral oophorectomy) alone without removal of the ovaries at the time of surgery. Furthermore, we will extend the collection to cells from the fallopian tubes in 225 women for a total population of 400.

We will administer a questionnaire assessing endometrial and ovarian cancer risk factors and gynecologic history; obtain blood and urine; and obtain carefully-mapped frozen and fixed endometrial and ovarian tissues. We will immunostain endometrial tissues to assess the presence, number, location, and size of foci containing PTEN-null glands, which represents a validated surrogate of mutations in the PTEN tumor suppressor gene. This pilot will demonstrate the feasibility of executing this complex protocol; determine the number and spacing of sections required to accurately and efficiently assess the PTEN status of the endometrium; and provide data for developing power estimates needed to propose a full-scale study with a sufficient number of subjects to test our hypothesis that PTEN abnormalities account for a substantial proportion of the risk associated with recognized epidemiologic endometrial cancer risk factors. It will assess the feasibility of performing molecular analyses on ovarian surface epithelial cells and tubal cells collected intra-operatively, and correlating molecular findings with known ovarian cancer risk factors. If successful, this will provide the basis for larger studies aimed at identifying early molecular events in

ovarian carcinogenesis, particularly in the setting of women at increased genetic

risk of ovarian cancer. The pilot itself will also provide an extremely valuable

repository for future biomarker pilot studies.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Inclusion criteria include: 18 years of age and older with:

  * a benign condition for which subject has decided to have a hysterectomy (removal of the uterus), performed through an abdominal incision (open procedure) or through a laparoscope (minimally invasive procedure). The hysterectomy can be performed with or without removal of the tubes, ovaries or cervix.
  * a benign cyst on the ovary(s) which subject has decided to have removed, with or without removal of the entire ovary. The surgery will be done with either an abdominal incision (open) or through a laparoscope (minimally invasive procedure).
  * positive test for the BRCA 1 or 2 gene, which puts subject at an increased risk for breast cancer, and subject has decided to undergo surgery (either with an abdominal incision or through a laparoscope) to remove the uterus, tubes and ovaries, or any combination
  * diagnosis of ovarian cancer or possible ovarian cancer and subject has been advised to undergo a hysterectomy (removal of the uterus), removal of the tubes and ovaries or any combination, with an abdominal incision or through a laparoscope.

EXCLUSION CRITERIA:

Evidence on gross examination of the surgically removed uterus that there is a carcinoma invading the myometrium; however, post-operative diagnosis of early endometrial carcinoma will not be a cause for post-hoc exclusion after specimen and data collection. We will exclude women with a previous gynecologic or gastrointestinal cancer. At the discretion of the surgeon, we will exclude women with cancer in whom the study procedures may interfere with clinical management (e.g. staging of the cancer). We will exclude women who had neo-adjuvant chemotherapy and women who underwent chemoprevention of ovarian or breast cancer. We will also exclude women currently wearing an intrauterine device.

Ages: 18 Years to 54 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women undergoing hysterectomy and/or unilateral or bilateral oophorectomy for benign indications, women at high risk or ovarian cancer or women with diagnosed ovarian cancer at Magee Women s Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 359 (Actual)
Dates: Start 2006-04-24 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-11-13 (Actual)

PRIMARY OUTCOMES:
Feasibility of sampling and recruiting | Ongoing
  Successful enrollment of women undergoing benign surgery, surgery because of high risk of ovarian cancer, or surgery because of diagnosed ovarian cancer.
Assessing PTEN abnormalities in benign tissue | Ongoing
  Histological assessment of PTEN staining in normal endometrial tissues.
Optimization of PTEN testing | Ongoing
  Improvement of PTEN staining after modifying the immunohistochemical staining protocol.
Feasibility of additional assays | Ongoing
  Pilot testing of other assays on tissue and cytology samples.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Wentzensen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Magee Women's hospital, Pittsburgh, Pennsylvania, United States